CLINICAL TRIAL: NCT02828371
Title: Effectiveness of a Very Early Stepping Verticalization Protocol in Severe Acquired Brain Injured Patients: a Randomized Pilot Study in ICU
Brief Title: Early Stepping Verticalization in ICU for ABI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Erigo_eff
Record Dates: First submitted 2016-07-02; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Brain Injury; Consciousness Disorders
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Erigo (Experimental): Single daily sessions of verticalization, using a tilt table with an integrated robotic stepping device (Erigo. Hocoma AG, Switzerland) located in the ICU room. Sessions were performed five times per week (Monday-Friday) for three consecutive weeks (a total of 15 sessions per patient). On the same days the patients received conventional physiotherapy for 30 minutes a day. Before the verticalization period the experimental group received conventional in-bed physiotherapy for 60 minutes a day.
  Interventions: Device: stepping verticalization
- Conventional (Active Comparator): treated with conventional in-bed physiotherapy for 60 minutes a day, from Monday to Friday, throughout the ICU stay.
  Interventions: Other: conventional mobilization

INTERVENTIONS:
Device: stepping verticalization — After patient positioning, the slope of the tilt table was gradually increased from 0° to 20°, 40° and then 60° in a time span of nine minutes. The stepping frequency was set at 20 steps/min for the entire treatment. Cardiovascular and respiratory parameters were continuously monitored. The net time of the session was 30 minutes
  Arms: Erigo
Other: conventional mobilization — in-bed physiotherapy (mobilization exercises in supine and sitting position on bed, without out-of-bed mobilization nor verticalization)
  Arms: Conventional

SUMMARY:
Verticalization was reported to improve the level of arousal and awareness in patients with severe acquired brain injury (ABI) and to be safe in ICU. The investigators evaluated the effectiveness of a very early stepping verticalization protocol on the functional and neurological outcome of patients affected by disorder of consciousness due to ABI.

Consecutive patients with Vegetative State or Minimally Conscious State were enrolled in ICU on the third day after an ABI. They were randomized to undergo conventional physiotherapy alone or associated to fifteen 30-minute sessions of verticalization, using a tilt table with robotic stepping device. Once stabilized, patients were transferred to a Neurorehabilitation unit for an individualized treatment. Outcome measures were assessed on the third day from the injury (T0), at ICU discharge (T1) and at Rehab discharge (T2).

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale (GCS) ≤8 for ≥24h from the event;
* diagnosis of vegetative state or minimally conscious state on the third day after the injury;
* adequate pulmonary gas exchanging function;
* stable hemodynamics

Exclusion Criteria:

* sedation;
* unstable intracranial pressure (ICP);
* cerebral perfusion pressure (CPP) <60 mmHg;
* fractures or skin lesions in thorax, abdomen or lower limbs;
* deep vein thrombosis;
* body weight >130 kg; height >210 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale change | through study completion, average 18 weeks
Glasgow Coma Scale change | through study completion, average 18 weeks
Levels of Cognitive Functioning change | through study completion, average 18 weeks
Disability Rating Scale change | through study completion, average 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona "Moriggia Pelascini", Gravedona Ed Uniti, CO, Italy

REFERENCES:
- [Derived] Frazzitta G, Zivi I, Valsecchi R, Bonini S, Maffia S, Molatore K, Sebastianelli L, Zarucchi A, Matteri D, Ercoli G, Maestri R, Saltuari L. Effectiveness of a Very Early Stepping Verticalization Protocol in Severe Acquired Brain Injured Patients: A Randomized Pilot Study in ICU. PLoS One. 2016 Jul 22;11(7):e0158030. doi: 10.1371/journal.pone.0158030. eCollection 2016. PMID 27447483